CLINICAL TRIAL: NCT02649608
Title: Interventional, Open-label, Exploratory Study Investigating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Lu AE04621 and the Active Metabolite Lu AA40326 After Ascending Oral Doses of Lu AE04621 to Patients With Parkinson's Disease
Brief Title: An Exploratory Study Investigating Safety, Tolerability and Pharmacokinetics of Ascending Doses of Lu AE04621 in Parkinson Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16779A
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study comprised 5 cohorts (Cohorts 1 to 5), with each cohort consisting of 3 patients (men and/or women). The dosing regimen planned for Cohort 1 was a dose of 0.2 mg Lu AE04621 on Day 1 followed by a dose of 0.4 mg Lu AE04621 on Day 2, and a dose of 0.6 mg Lu AE04621 on Day 3. • The dosing regimen planned for Cohort 2 was 0.4 mg Lu AE04621 on Day 1 followed by a dose of 0.6 mg Lu AE04621 on Day 2, and a dose of 0.8 mg Lu AE04621 on Day 3. The dosing regimen planned for Cohort 3 was 0.2 mg Lu AE04621 on Day 1 followed by a dose of 0.4 mg Lu AE04621 on Day 2, a dose of 0.6 mg Lu AE04621 on Day 3, and a dose of 1.0 mg Lu AE04621 on Day 4. The dosing regimen planned for Cohorts 4 and 5 was 0.2 mg Lu AE04621 on Day 1 followed by a dose of 0.4 mg Lu AE04621 on Day 2, a dose of 0.6 mg Lu AE04621 on Day 3, and a dose of 1.2 mg Lu AE04621 on Day 4. The results are presented by dose groups and are based on the actual doses administered.
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 0.04 mg Lu AE04621 (Experimental): Patients having received a dose of 0.04 mg, independent of which Cohort they belong to.
  Interventions: Drug: 0.04 mg Lu AE04621
- 0.08 mg Lu AE04621 (Experimental): Patients having received a dose of 0.08 mg, independent of which Cohort they belong to.
  Interventions: Drug: 0.08 mg Lu AE04621
- 0.2 mg Lu AE04621 (Experimental): Patients having received a dose of 0.2 mg, independent of which Cohort they belong to.
  Interventions: Drug: 0.2 mg Lu AE04621
- 0.4 mg Lu AE04621 (Experimental): Patients having received a dose of 1.2 mg, independent of which Cohort they belong to.
  Interventions: Drug: 0.4 mg Lu AE04621
- 0.6 mg Lu AE04621 (Experimental): Patients having received a dose of 0.6 mg, independent of which Cohort they belong to.
  Interventions: Drug: 0.6 mg Lu AE04621
- 0.8 mg Lu AE04621 (Experimental): Patients having received a dose of 0.8 mg, independent of which Cohort they belong to.
  Interventions: Drug: 0.8 mg Lu AE04621
- 1.0 mg Lu AE04621 (Experimental): Patients having received a dose of 1.0 mg, independent of which Cohort they belong to.
  Interventions: Drug: 1.0 mg Lu AE04621
- 1.2 mg Lu AE04621 (Experimental): Patients having received a dose of 1.2 mg, independent of which Cohort they belong to.
  Interventions: Drug: 1.2 mg Lu AE04621

INTERVENTIONS:
Drug: 0.04 mg Lu AE04621 — 0.04 mg dose group
  Arms: 0.04 mg Lu AE04621
Drug: 0.08 mg Lu AE04621 — 0.08mg dose group
  Arms: 0.08 mg Lu AE04621
Drug: 0.2 mg Lu AE04621 — 0.2 mg dose group
  Arms: 0.2 mg Lu AE04621
Drug: 0.4 mg Lu AE04621 — 0.4 mg dose group
  Arms: 0.4 mg Lu AE04621
Drug: 0.6 mg Lu AE04621 — 0.6 mg dose group
  Arms: 0.6 mg Lu AE04621
Drug: 0.8 mg Lu AE04621 — 0.8 mg dose group
  Arms: 0.8 mg Lu AE04621
Drug: 1.0 mg Lu AE04621 — 1.0 mg dose group
  Arms: 1.0 mg Lu AE04621
Drug: 1.2 mg Lu AE04621 — 1.2 mg dose group
  Arms: 1.2 mg Lu AE04621

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics, and efficacy of the Lu AE04621 and metabolite after ascending oral doses of Lu AE04621 in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
The study comprised 5 cohorts (Cohorts 1 to 5), with each cohort consisting of 3 patients with Parkinson's disease (men and/or women). Each patient will be treated for 3 or 4 days, with increasing dose each day.

Dosing regimen will be decided at a dosing conferences. Dose levels can be increased, maintained or reduced both between cohorts but also within same cohort. The results are presented by dose level and reflect the actual doses administered.

A follow-up safety visit was scheduled approximately 7 days after the last dose of IMP.

ELIGIBILITY:
Inclusion Criteria:

* The patient is diagnosed with idiopathic Parkinson Disease (consistent with the UK Parkinson's Disease Society Brain Bank Criteria for the Diagnosis of PD).
* The patient's Hoehn and Yahr Staging score is ≤ 3 in the "ON" state.
* The patient experiences motor fluctuations with at least 2.5 hours of "OFF" periods in the awake time and has predictable morning "OFF" episodes, which have been consistent within the past 4 weeks.
* The patient currently has a good response to L-DOPA and has been receiving a stable dose of L-DOPA (≥3 doses per day of standard L-DOPA or ≥3 doses per day of Carbidopa and L-DOPA, Extended-Release Capsules) during at least four weeks prior to screening.

Exclusion Criteria:

* The patient has cognitive impairment, defined as a Mini Mental State Examination(MMSE) score ≤ 26 at the Screening Visit.
* The patient has severe disabling dyskinesia
* The patient takes or has taken disallowed recent or concomitant medication (CYP2D6 inhibitors, CYP 3A4 substrate, Dopamine agonists, 5 HT3 antagonists, Anti-viral (Amantadine))

Other protocol defined inclusion and exclusion criteria may apply

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (4):
- United States (4):
  - US1251, Hallandale, Florida
  - US1126, Orlando, Florida
  - US1352, Chicago, Illinois
  - US1084, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Groups are overlapping the cohorts
Groups:
- Group 1: Patients received 0.2 mg, 0.4 mg, and 0.6 mg Lu AE04621 on Days 1, 2, and 3, respectively
- Group 2: Patient received 0.2 mg, 0.4 mg, and 0.2 mg Lu AE04621 on Days 1, 2, and 3, respectively
- Group 3: Patients received 0.4 mg, 0.6 mg, and 0.8 mg Lu AE04621 on Days 1, 2, and 3, respectively
- Group 4: Patients received 0.2 mg, 0.4 mg, 0.6 mg, and 1.0 mg Lu AE04621 on Days 1, 2, 3, and 4, respectively
- Group 5: Patients received 0.2 mg, 0.4 mg, 0.6 mg, and 1.2 mg Lu AE04621 on Days 1, 2, 3, and 4, respectively
- Group 6: Patients received 0.2 mg, 0.4 mg, 0.4 mg, and 0.4 mg Lu AE04621 on Days 1, 2, 3, and 4, respectively
- Group 7: Patient received 0.04 mg, 0.08 mg, 0.6 mg, and 0.6 mg Lu AE04621 on Days 1, 2, 3, and 4, respectively
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Started | 2 | 1 | 3 | 3 | 3 | 2 | 1
Completed | 2 | 1 | 3 | 3 | 3 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total patient population
Groups:
- Lu AE04621: Patients having received 3 or 4 doses of Lu AE04621, ranging from 0.04 to 1.2 mg. Baseline measures are anlayzed on full patient group only.
Arm/Group | Lu AE04621
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Based on the Safety Variables (Adverse Events, Clinical Safety Laboratory Tests, Vital Signs, Weight, and ECG)
Description: Number of patients with an adverse event
Time Frame: Baseline to day 11
Population: Each patient received 3 or 4 doses of Lu AE04621. The overall number of participants analyzed in each group represents the number of patients having received a particular dose.
Measure: Count of Participants; unit: Participants
Groups:
- 0.4 mg Lu AE04621: Patients having received a dose of 0.4 mg, independent of which Cohort they belong to
Arm/Group | 0.04 mg Lu AE04621 | 0.08 mg Lu AE04621 | 0.2 mg Lu AE04621 | 0.4 mg Lu AE04621 | 0.6 mg Lu AE04621 | 0.8 mg Lu AE04621 | 1.0 mg Lu AE04621 | 1.2 mg Lu AE04621
Number analyzed (Participants) | 1 | 1 | 11 | 14 | 12 | 3 | 3 | 3
Participants | 0 | 0 | 2 | 7 | 3 | 3 | 1 | 1

2. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC(0-24 Hours)) for Lu AE04621
Time Frame: From dosing to up to 24 hours after dosing
Population: The overall number of participants analyzed in each group represents the number of dosing occasion at a particular dose, minus occasions with missing or unreliable data. The results are reported for the dose groups with sufficient data to calculate the parameter (missing dose groups for AUC(0-24 hours) are: 0.04, 0.08, 0.8, 1.0 and 1.2 mg)
Measure: Mean (Standard Deviation); unit: pgxh/mL
Groups:
- 0.4 mg Lu AE04621: Patients having received a dose of 0.4 mg Lu AE04621, independent of which cohort they belong to.
- 0.6 mg Lu AE04621: Patients having received a dose of 0.6 mg Lu AE04621, independent of which cohort they belong to.
Arm/Group | 0.2 mg Lu AE04621 | 0.4 mg Lu AE04621 | 0.6 mg Lu AE04621
Number analyzed (Participants) | 9 | 11 | 9
pgxh/mL | 212 (268) | 292 (219) | 309 (276)

3. Primary Outcome: Maximum Observed Concentration (Cmax) for Lu AE04621
Time Frame: From dosing to up to 24 hours after dosing
Population: Each patient received 3 or 4 doses of Lu AE04621. The overall number of participants analyzed in each group represents the number of dosing occasion at a particular dose, minus occasions with missing or unreliable data.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- 0.08 mg LuAE04621: Patients having received a dose of 0.08 mg, independent of which Cohort they belong to.
- 0.6 mg Lu AE06421: Patients having received a dose of 0.6 mg, independent of which Cohort they belong to.
Arm/Group | 0.04 mg Lu AE04621 | 0.08 mg LuAE04621 | 0.2 mg Lu AE04621 | 0.4 mg Lu AE04621 | 0.6 mg Lu AE06421 | 0.8 mg Lu AE04621 | 1.0 mg Lu AE04621 | 1.2 mg Lu AE04621
Number analyzed (Participants) | 1 | 1 | 11 | 17 | 13 | 2 | 3 | 2
pg/mL | 3.52 (0) | 6.31 (0) | 48.6 (69.9) | 60.4 (57.3) | 52.8 (48.5) | 29.8 (31.3) | 55.9 (60.7) | 237 (67.9)

4. Primary Outcome: Apparent Elimination Half-life of Lu AE04621 in Plasma (t½)
Time Frame: From dosing to up to 24 hours after dosing
Population: The overall number of participants analyzed in each group represents the number of dosing occasion at a particular dose, minus occasions with missing or unreliable data. The results are reported for the dose groups with sufficient data to calculate the parameter (missing dose groups for t½ are: 0.04, 0.08, 0.8, 1.0 and 1.2 mg)
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 0.2 mg Lu AE04621 | 0.4 mg Lu AE04621 | 0.6 mg Lu AE04621
Number analyzed (Participants) | 9 | 10 | 9
hour | 3.24 (2.43) | 5.00 (2.51) | 4.11 (2.01)

5. Primary Outcome: Time to Onset of "ON" Time After Lu AE04621 Administration
Description: "ON" state is defined as a period of good control of parkinsonian features with relatively good overall function and mobility. Motor fluctuation assessments are patient-reported outcomes, and guidance will be given to the patients on how to complete them. Date and time will be registered when the patient turns to "ON" and "OFF" state. "OFF" state is defined as a period of poor control of parkinsonian features with relatively poor overall function, such as worsening tremor, rigidity, balance or bradykinesia.
  Data are no presented for the dose groups 0.04, 0.08, and 1.0 mg Lu AE04621 since no patients turned 'ON'.
Time Frame: From dosing to 90 minutes after dosing
Population: Each patient received 3 or 4 doses of Lu AE04621. The overall number of participants analyzed in each group represents the number of dosing occasion at a particular dose. Data are no presented for the dose groups 0.04, 0.08, and 1.0 mg Lu AE04621 since no patients turned 'ON'.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: dosing occasion when patient turned ON
Arm/Group | 0.2 mg Lu AE04621 | 0.4 mg Lu AE04621 | 0.6 mg Lu AE04621 | 0.8 mg Lu AE04621 | 1.2 mg Lu AE04621
Number analyzed (Participants) | 12 | 18 | 13 | 3 | 3
Number analyzed (dosing occasion when patient turned ON) | 6 | 11 | 7 | 1 | 2
minutes | 35 (20.4) | 41 (28.6) | 39 (22.7) | 17 (0) | 20 (17)

6. Primary Outcome: Duration of "ON" Time
Description: "ON" state is defined as a period of good control of parkinsonian features with relatively good overall function and mobility. Motor fluctuation assessments are patient-reported outcomes, and guidance will be given to the patients on how to complete them. Date and time will be registered when the patient turns to "ON" and "OFF" state. "OFF" state is defined as a period of poor control of parkinsonian features with relatively poor overall function, such as worsening tremor, rigidity, balance or bradykinesia. Outcome measured in minutes.
  Data are no presented for the dose groups 0.04, 0.08, and 1.0 mg Lu AE04621 since no patients turned 'ON' following administration of Lu AE04621.
Time Frame: From dosing up to 24h post-dose
Population: Each patient received 3 or 4 doses of Lu AE04621. The overall number analyzed in each group represents the number of dosing occasion at a particular dose when patients turned 'ON'. Data are no presented for the dose groups 0.04, 0.08, and 1.0 mg Lu AE04621 since no patients turned 'ON'.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 0.2 mg Lu AE04621 | 0.4 mg Lu AE04621 | 0.6 mg Lu AE06421 | 0.8 mg Lu AE04621 | 1.2 mg Lu AE04621
Number analyzed (Participants) | 6 | 11 | 7 | 1 | 2
minutes | 203 (152.9) | 249 (98.9) | 270 (124.7) | 87 (0) | 401 (209.3)

ADVERSE EVENTS:
Time Frame: Baseline to day 11
Description: Treatment-emergent adverse events are reported in this section.
Arm/Group | 0.04 mg Lu AE04621 | 0.08 mg Lu AE04621 | 0.2 mg Lu AE04621 | 0.4 mg Lu AE04621 | 0.6 mg Lu AE04621 | 0.8 mg Lu AE04621 | 1 mg Lu AE04621 | 1.2 mg Lu AE04621
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/11 | 0/14 | 0/12 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/11 | 0/14 | 0/12 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 2/11 | 7/14 | 3/12 | 3/3 | 1/3 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.04 mg Lu AE04621 (N=1) | 0.08 mg Lu AE04621 (N=1) | 0.2 mg Lu AE04621 (N=11) | 0.4 mg Lu AE04621 (N=14) | 0.6 mg Lu AE04621 (N=12) | 0.8 mg Lu AE04621 (N=3) | 1 mg Lu AE04621 (N=3) | 1.2 mg Lu AE04621 (N=3)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Blunted affect (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Because of the limit of quantification, some missing and/or unreliable data prevented the calculation of some of the PK parameters (AUC0-24hours, apparent elimination half-life) for some of the dose groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes